CLINICAL TRIAL: NCT00444392
Title: Impact of Gastric Bypass Surgery on Risk of CVD in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 061003; 1K23DK075907-01 (NIH)
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Obese Patients; Type 2 Diabetes Mellitus
Keywords: Obese; type 2 Diabetes Mellitus; Gastric Bypass Surgery; Risk of CVD
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Calorie controlled diabetic diet for the control patients — Calorie controlled diabetic diet for the control patients

SUMMARY:
Central hypothesis is: Gastric bypass surgery reduces the risk of CVD in morbidly obese subjects (defined as BMI ≥35 kg/m2) with T2DM.

To determine whether surgically induced weight loss decreases the risk of CVD in morbidly obese subjects with T2DM. I hypothesize that patients with T2DM who undergo gastric bypass surgery will significantly reduce mean levels of risk factors for CVD compared with diabetic individuals with the same BMI who maintain their weight.

DETAILED DESCRIPTION:
Patients with type 2 diabetes mellitus (T2DM) are more likely to die from cardiovascular diseases (CVD) than people without diabetes. Furthermore, patients with diabetes have not benefited from the advances in the management of CVD and/or its risk factors that have resulted in a decrease in mortality for CVD patients without diabetes. Short-term studies have demonstrated that weight loss in overweight or obese subjects with T2DM is associated with decreased insulin resistance, substantial improvements in glycemic and lipoprotein profile, and reduction in blood pressure. However, long-term data substantiating that these improvements can be maintained are limited. Obesity, and susceptibility to weight gain, is a chronic condition. Continuous care is required to avoid weight regain especially after intensive weight loss. Morbidly obese patients with body mass index (BMI) over 35 kg/m2 have significant difficulty maintaining weight loss adequate to resolve obesity-related medical conditions by changes in lifestyle or pharmacologic strategies. Currently, surgical treatment of morbid obesity, termed bariatric surgery, appears to be the only modality that results in significant and sustained weight loss along with reversal of diabetes and improvements in cholesterol biosynthesis, and lipoprotein metabolism in morbidly obese patients. Given these observations, we question if patients with T2DM who undergo gastric bypass surgery will significantly reduce levels of abnormalities in vascular structure and function that are central to the development of atherosclerosis. In Specific Aim 1, we will determine whether surgically induced weight loss decreases the risk of CVD in morbidly obese subjects with T2DM. In Specific Aim 2, we will elucidate the mechanisms by which surgically induced weight loss reduces over time the risk of CVD in morbidly obese subjects with T2DM. The proposed study is a prospective cohort clinical trial aimed to evaluate changes over time in cardiovascular structure and function of morbidly obese subjects with T2DM undergoing gastric bypass surgery compared to a matched control group who do not undergo gastric bypass surgery. The results of the proposed studies will provide the foundation for a new clinical strategy aimed to prevent the development of CVD in obese patients with T2DM. Furthermore, they will serve as the baseline for future large scale longitudinal studies based on aggregate occurrence of severe cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of T2DM diabetes mellitus with HbA1c ≤ 10.0%

   Any one of the following will be considered to be sufficient evidence that diabetes is present:
   * Current regular use of insulin
   * Current regular use of oral hypoglycemic medication.
   * Documented diabetes by current ADA criteria (98).
2. Body mass index ≥ 35 kg/m2 in accord with the 1991 NIH obesity surgery consensus conference criteria and stable weight for the previous 3 months (99).
3. Age between 18-60 years old. Individuals older than 60 years of age are excluded due to their increased risk of mortality and peri-operative morbidity.
4. Ability and willingness to provide informed consent.
5. No expectation that subject will be moving out of the area of the clinical center during the next 24 months.

Exclusion Criteria:

1. Presence of CVD defined as: CAD, electrocardiographic criteria for past myocardial infarction(s), ischemic stroke, peripheral artery bypass surgery, percutaneous transluminal angioplasty, or amputation because of atherosclerotic disease.
2. Significant non-diabetic co-morbidity affecting life expectancy (e.g., malignancy).
3. Significant other co-morbidities (e.g. psychiatric disorder) that results in ineligibility for gastric bypass surgery.
4. Pregnancy or planning pregnancy.
5. Severe dyslipidemia (triglycerides >600 mg/dl or cholesterol >350 mg/dl).
6. Uncontrolled hypertension.
7. Smoking.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Carotid artery intima-media thickness | 6 month, 1 year
Brachial artery flow mediated dilation | 6 month, 1 year

SECONDARY OUTCOMES:
Insulin Sensitivity | 6 month, 1 year
Body Composition | 6 month, 1 year
Lipoprotein Profiles | 6 months, 1 year
Inflammatory Markers | 6 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Torquati, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States